# Statistical Analysis Plan J2X-MC-PYAG

A Randomized, Placebo-Controlled, Participant- and Investigator-Blind, Phase 1 Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of LY3819253 Administered Subcutaneously to Healthy Participants

NCT04537910

Approval Date: 01-Sep-2020

# STATISTICAL ANALYSIS PLAN

A Randomized, Placebo-Controlled, Participant- and Investigator-Blind, Phase 1 Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of LY3819253 Administered Subcutaneously to Healthy Participants

Statistical Analysis Plan Status: Final Statistical Analysis Plan Date: 28 August 2020

Study Drug: LY3819253

Sponsor Reference: J2X-MC-PYAG Covance CRU Study: 1000071-8450508

Clinical Phase I

Approval Date: 01-Sep-2020 GMT

Final, 28 August 2020 

# 1. TABLE OF CONTENTS

| 1. | TABLE | OF CONTENTS | 2 |
|-----------|---------|-------------------------------------------------|----|
| 2. | ABBRE | EVIATIONS | 4 |
| 3. | INTRO | DUCTION | 6 |
| 4. | STUDY | OBJECTIVES AND ENDPOINTS | 6 |
| <b>5.</b> | STUDY | DESIGN | 7 |
| | 5.1 Ove | erall Design | 7 |
| | 5.2 Scr | eening and Enrollment | 7 |
| | 5.3 Inp | atient Stay | 7 |
| | 5.4 Out | patient Follow-up | 8 |
| 6. | TREAT | MENTS | 8 |
| 7. | SAMPI | E SIZE JUSTIFICATION | 9 |
| 8. | DEFIN | TION OF ANALYSIS POPULATIONS | 9 |
| 9. | STATIS | STICAL METHODOLOGY | 9 |
| | 9.1 Ger | neral | 9 |
| | 9.2 Dei | nographics and Subject Disposition | 10 |
| | 9.3 Pha | rmacokinetic Assessment | 10 |
| | 9.3.1 | Pharmacokinetic Analysis | 10 |
| | 9.3.2 | Pharmacokinetic Statistical Methodology | 14 |
| | 9.4 Saf | ety and Tolerability Assessments | 15 |
| | 9.4.1 | Adverse events | 15 |
| | 9.4.2 | Concomitant medication | 15 |
| | 9.4.3 | Clinical laboratory parameters | 15 |
| | 9.4.4 | Vital signs | 16 |
| | 9.4.5 | Electrocardiogram (ECG) | 16 |
| | 9.4.6 | Immunogenicity Assessments | 16 |
| | 9.4.7 | Injection-Site Reactions | 16 |
| | 9.4.8 | Visual Analog Scale (VAS) Analysis | 16 |
| | 9.4.9 | Hypersensitivity reactions | |
| | 9.4.10 | Other assessments | 16 |
| | 9 4 11 | Safety and Tolerability Statistical Methodology | 17 |

# $\begin{cal}CONFIDENTIAL\\Sponsor Reference J2X-MC-PYAG\end{cal}$

| 10. | INTERIM ANALYSES | .17 |
|------------|----------------------------------------------------------|-----|
| 11. | CHANGES FROM THE PROTOCOL SPECIFIED STATISTICAL ANALYSES | .17 |
| <b>12.</b> | REFERENCES | .17 |
| 13. | DATA PRESENTATION | .17 |
| | 13.1 Derived Parameters | .17 |
| | 13.2 Missing Data | .17 |
| | 13.3 Insufficient Data for Presentation | |

Final, 28 August 2020 

#### 2. ABBREVIATIONS

Abbreviations pertain to the Statistical Analysis Plan (SAP) only (not the tables, figures and listings [TFLs]).

%AUC( $t_{last}$ - $\infty$ ) Percentage of AUC(0- $\infty$ ) extrapolated

ADA Antidrug antibody

AE Adverse event

AUC Area under the concentration versus time curve

 $AUC(0-\infty)$  Area under the concentration versus time curve from time zero to infinity

 $AUC(0-t_{last})$  Area under the concentration versus time curve from time zero to time t,

where t is the last time point with a measurable concentration

BQL Below the lower limit of quantitation

CL/F Apparent total body clearance of drug calculated after extra-vascular

administration

C<sub>max</sub> Maximum observed drug concentration

CRF Case Report Form

CRU Clinical Research Unit
CSR Clinical Study Report

CV Coefficient of variation

ECG Electrocardiogram

ICH International Conference on Harmonisation

ISR Injection-site reaction

MedDRA Medical Dictionary for Regulatory Activities

PK Pharmacokinetic

SAE Serious adverse event
SAP Statistical Analysis Plan

SARS-COV-2 Severe acute respiratory syndrome coronavirus 2

SC Subcutaneous

SD Standard deviation

 $t_{1/2}$  Half-life associated with the terminal rate constant  $(\lambda_z)$  in non-

compartmental analysis

TE ADA Treatment-emergent antidrug antibodies

TEAE Treatment-emergent adverse event

Final, 28 August 2020 

| TFLs | Tables, Figures, and Listings |
|---|---|
| $t_{max}$ | Time of maximum observed drug concentration |
| VAS | Visual analog scale |
| $V_z/F$ | Apparent volume of distribution during the terminal phase after extravascular administration |
| WHO | World Health Organization |

Final, 28 August 2020 

# 3. INTRODUCTION

This SAP has been developed after review of the Clinical Study Protocol (final version dated 17 August 2020).

This SAP describes the planned analysis of the safety, tolerability and pharmacokinetic (PK) data from this study. A detailed description of the planned TFLs to be presented in the clinical study report (CSR) is provided in the accompanying TFL shell document.

The intent of this document is to provide guidance for the statistical and PK analyses of data. In general, the analyses are based on information from the protocol, unless they have been modified by agreement with Eli Lilly and Company. A limited amount of information concerning this study (e.g., objectives, study design) is given to help the reader's interpretation. When the SAP and TFL shells are agreed upon and finalized, they will serve as the template for this study's CSR.

This SAP supersedes the statistical considerations identified in the protocol; where considerations are substantially different, they will be so identified. If additional analyses are required to supplement the planned analyses described in this SAP, they may be performed and will be identified in the CSR. Any substantial deviations from this SAP will be agreed upon with Eli Lilly and Company and identified in the CSR. Any minor deviations from the TFLs may not be documented in the CSR.

This SAP is written with consideration of the recommendations outlined in the International Conference on Harmonisation (ICH) E9 Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials<sup>1</sup> and the ICH E3 Guideline entitled Guidance for Industry: Structure and Content of Clinical Study Reports<sup>2</sup>.

# 4. STUDY OBJECTIVES AND ENDPOINTS

| Objectives | Endpoints |
|---|---|
| Primary To determine the PK of single subcutaneous (SC) doses of LY3819253 in healthy participants | Area under the concentration versus time curve from time zero to infinity $(AUC(0-\infty))$ |
| Secondary To describe safety and tolerability following single SC doses of LY3819253 in healthy participants | Incidence of spontaneously reported adverse events (AEs), treatment-emergent adverse events (TEAEs), and serious adverse events (SAEs); vital signs; clinical laboratory results |
| Exploratory To assess injection-site reactions (ISRs) following single SC doses of LY3819253 in healthy participants | Characterization and measurement of incidence and severity of ISRs, including injection site pain, using data collected from the ISR assessment, as well as the exploratory tool (Scarletred). |

Final, 28 August 2020 

| To determine the immunogenicity of | Incidence of treatment-emergent antidrug |
|---|---|
| LY3819253 following single SC doses in | antibodies (TE ADA). |
| healthy participants. | |

#### 5. STUDY DESIGN

# 5.1 Overall Design

This is a single-site study in healthy participants who will receive a single SC dose of LY3819253. The study will be participant- and investigator-blinded, randomized, and placebo controlled. A study schema for this study can be seen in Figure 1.



Abbreviations: LY = LY3819253; PBO = placebo; SC = subcutaneous.

Figure 1: Study Schema for Study J2X-MC-PYAG

# 5.2 Screening and Enrollment

Up to 3 cohorts may be enrolled with at least 9 participants per cohort (7 LY3819253: 2 placebo), with the intention that at least 6 participants randomized to LY3819253 have sufficient evaluable data in each cohort.

Participants will be screened within 14 days prior to Day 1 of dosing for each cohort. Participants will be admitted to the clinical research unit (CRU) as part of an inpatient visit on Day -1 and will be sequentially enrolled and then randomized to treatment.

# 5.3 Inpatient Stay

Participants will be admitted to the study site on Day -1. They will remain inpatient until discharge on Day 7 after study procedures are complete.

Final, 28 August 2020 

#### **Dosing**

Dosing will occur on Day 1. Intended doses of LY3819253 are as follows:

- Cohort 1: 350 mgCohort 2: 700 mg
- Cohort 3 (optional): 700 mg (alternative injection volumes)

Participants will undergo PK sampling and safety assessment after dosing.

For Cohorts 1 and 2, a safety review will be conducted to determine whether it is appropriate to proceed with dosing of the next cohort. This safety review will be conducted based on data from at least 4 participants, after at least 4 days after dosing.

# **Sentinel dosing**

Cohort 1 will include sentinel dosing. The first 2 participants will be randomized and dosed (1 LY3819253: 1 placebo).

The investigator and the Lilly sponsor team are responsible for determining if safety and tolerability is acceptable to continue with dosing subsequent participants.

Tolerability as measured by ISRs and their severity is anticipated to be the main safety consideration for this assessment. While no serious systemic reactions have been seen with LY3819253 to date, participants will be closely monitored.

If the investigator and Lilly sponsor team determine that safety and tolerability is acceptable, the remaining participants in the cohort will be dosed on the next day.

Cohort 2 and the optional Cohort 3 will not include sentinel dosing.

# Postdose sampling

On Days 1 through 7, participants will undergo PK sampling and safety assessment.

# 5.4 Outpatient Follow-up

Follow-up visits will be conducted through Day 85.

In the event a participant has suspected or confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, follow-up visits may be conducted at the participant's home.

#### 6. TREATMENTS

The following is a list of the study treatment abbreviations that will be used in the TFLs.

Final, 28 August 2020 

| Cohort | Study Treatment Name* | Treatment order in TFL |
|---|---|---|
| All | Placebo SC | 1 |
| 1 | 350 mg LY3819253 SC (2x 1.4 mL) | 2 |
| 2 | 700 mg LY3819253 SC (1x 1.4 mL + 2x 2.1 mL) | 3 |
| 3 (optional) | 700 mg LY3819253 SC (1x1.8 mL + 2x 1.9 mL) | 4 |

<sup>\*</sup>The LY3819253 formulation concentration will be 125 mg/mL in all cases.

#### 7. SAMPLE SIZE JUSTIFICATION

A maximum of 36 participants will be enrolled to study intervention with the intention that at least 6 participants randomized to LY3819253 have sufficient evaluable data in each cohort.

This would mean at least 12 participants with evaluable data if Cohorts 1 and 2 only are enrolled, or 18 participants if the optional Cohort 3 is also enrolled.

The sample size is not powered on the basis of statistical hypothesis testing. However, based on an assumption of 40% coefficient of variation (CV) for between subject variability in a PK parameter of interest, 6 subjects on active treatment per cohort may provide approximately 70% chance to ensure that a PK parameter's 90% confidence interval (CI) falls within (0.7, 1.43) over the corresponding geometric mean, such as  $AUC(0-\infty)$ .

A participant will be considered evaluable when the participant completes up to 29 days of study procedures. When a participant does not complete up to 29 days of study procedures, the sponsor will be consulted if the participant will need to be replaced.

#### 8. DEFINITION OF ANALYSIS POPULATIONS

The "Safety" population will consist of all participants who were randomly assigned and who received study intervention (LY3819253 or placebo). Participants will be analyzed according to the intervention they actually received.

The "Pharmacokinetic" population will consist of all treated participants who received study intervention (LY3819253) and have sufficient evaluable PK samples.

All protocol deviations that occur during the study will be considered for their severity/impact and will be taken into consideration when subjects are assigned to analysis populations.

#### 9. STATISTICAL METHODOLOGY

#### 9.1 General

Data listings will be provided for all data that is databased. Summary statistics and statistical analysis will only be presented for data where detailed in this SAP. For continuous data, summary statistics will include the arithmetic mean, arithmetic standard deviation (SD), median, minimum, maximum and N; for log-normal data (e.g. the PK parameters: area under the concentration versus time curve [AUCs] and maximum observed drug concentration [ $C_{max}$ ]) the geometric mean and geometric CV will also be presented. For categorical data, frequency count and percentages will be presented. Data listings will be provided for all subjects up to the point of withdrawal, with any subjects excluded from the relevant population highlighted. Summary

Final, 28 August 2020 

statistics and statistical analyses will generally only be performed for subjects included in the relevant analysis population. For the calculation of summary statistics and statistical analysis, unrounded data will be used.

Mean change from baseline is the mean of all individual subjects' change from baseline values. Each individual change from baseline will be calculated by subtracting the individual subject's baseline value from the value at the timepoint. The individual subject's change from baseline values will be used to calculate the mean change from baseline using a SAS procedure such as Proc Univariate.

Data analysis will be performed using SAS® Version 9.4 or greater.

# 9.2 Demographics and Subject Disposition

Subject disposition will be listed. The demographic variables age, sex, race, ethnicity, body weight, height and body mass index will be summarized and listed. All other demographic variables will be listed only.

#### 9.3 Pharmacokinetic Assessment

# 9.3.1 Pharmacokinetic Analysis

Noncompartmental methods applied with a validated software program, Phoenix WinNonlin (Certara, Version 8.1 or later) to the serum concentrations of LY3819253 will be used to determine the following PK parameters, when possible:

Final, 28 August 2020 

| Parameter | Units | Definition |
|---|---|---|
| $\overline{\mathrm{AUC}(0\text{-}\infty)}$ | μg*h/mL | area under the concentration versus time curve from time zero to infinity |
| $\%AUC(t_{last}-\infty)$ | % | percentage of AUC(0-∞) extrapolated |
| $AUC(0\text{-}t_{last})$ | μg*h/mL | area under the concentration versus time curve from time zero to time t, where t is the last time point with a measurable concentration |
| $C_{max}^{a}$ | $\mu g/mL$ | maximum observed drug concentration |
| $t_{max}$ | h | time of maximum observed drug concentration |
| t <sub>1/2</sub> | h | half-life associated with the terminal rate constant $(\lambda_z)$ in non-compartmental analysis |
| CL/F | L/h | apparent total body clearance of drug calculated after extra-vascular administration |
| V <sub>Z</sub> /F | L | apparent volume of distribution during the terminal phase after extra-vascular administration |

<sup>&</sup>lt;sup>a</sup> Serum LY3819253 drug concentration units will come in from the bioanalytical lab as ng/mL to one decimal place; the data will be transformed (unrounded) to  $\mu$ g/mL for analysis and reporting.

Additional PK parameters may be calculated, as appropriate. The software and version used for the final analyses will be specified in the CSR. Any exceptions or special handling of data will be clearly documented within the final study report.

Formatting of tables, figures and abbreviations will follow the Eli Lilly Global PK/PD/TS Tool: NON-COMPARTMENTAL PHARMACOKINETIC STYLE GUIDE. The version of the tool effective at the time of PK analysis will be followed.

#### **General PK Parameter Rules**

- Actual sampling times will be used in the final analyses of individual PK parameters, except for non-bolus pre-dose sampling times which will be set to zero.
- $C_{max}$  and  $t_{max}$  will be reported from observed values. If  $C_{max}$  occurs at more than one timepoint,  $t_{max}$  will be assigned to the first occurrence of  $C_{max}$ .
- AUC parameters will be calculated using a combination of the linear and logarithmic trapezoidal methods (linear-log trapezoidal rule). The linear trapezoidal method will be applied up to t<sub>max</sub> and then the logarithmic trapezoidal method will be used after t<sub>max</sub>. The minimum requirement for the calculation of AUC will be the inclusion of at least three consecutive serum concentrations above the lower limit of quantification, with at least one of these concentrations following C<sub>max</sub>. AUC(0-∞) values where the percentage of the total area extrapolated is more than 20% will be flagged. Any AUC(0-∞) value excluded from summary statistics will be noted in the footnote of the summary table.
- Half-life associated with the terminal rate constant ( $\lambda z$ ) in non-compartmental analysis ( $t_{1/2}$ ) will be calculated, when appropriate, based on the apparent terminal log-linear

Final, 28 August 2020 

portion of the concentration-time curve. The start of the terminal elimination phase for each subject will be defined by visual inspection and generally will be the first point at which there is no systematic deviation from the log-linear decline in serum concentrations. Half-life will only be calculated when a reliable estimate for this parameter can be obtained comprising of at least 3 data points. If  $t_{1/2}$  is estimated over a time window of less than 2 half-lives, the values will be flagged in the data listings. Any  $t_{1/2}$  value excluded from summary statistics will be documented in the footnote of the summary table.

- A uniform weighting scheme will be used in the regression analysis of the terminal loglinear portion of the concentration-time curve.
- The parameters based on predicted last quantifiable drug concentration will be reported.

#### **Individual PK Parameter Rules**

- Only quantifiable concentrations will be used to calculate PK parameters with the exception of special handling of certain concentrations reported below the lower limit of quantitation (BQL). Serum concentrations reported as BQL will be set to a value of zero when all of the following conditions are met:
  - o The compound is non-endogenous.
  - The samples are from the initial dose period for a subject or from a subsequent dose period following a suitable wash-out period.
  - The time points occur before the first quantifiable concentration.
- All other BQL concentrations that do not meet the above criteria will be set to missing.
- Also, where two or more consecutive concentrations are BQL towards the end of a profile, the profile will be deemed to have terminated and therefore any further quantifiable concentrations will be set to missing for the calculation of the PK parameters unless it is considered to be a true characteristic of the profile of the drug.

#### **Individual Concentration vs. Time Profiles**

- Individual concentrations will be plotted utilizing actual sampling times.
- The terminal point selections will be indicated on a semi-logarithmic plot.

# **Average Concentration vs. Time Profiles**

• The average concentration profiles will be graphed using scheduled (nominal) sampling times.

Final, 28 August 2020 

- The average concentration profiles will be graphed using arithmetic average concentrations.
- The pre-dose average concentration for single-dose data from non-endogenous compounds will be set to zero. Otherwise, only quantifiable concentrations will be used to calculate average concentrations.
- Concentrations at a sampling time exceeding the sampling time window specified in the protocol, or  $\pm$  10%, will be excluded from the average concentration profiles.
- Concentrations excluded from the mean calculation will be documented in the final study report.
- A concentration average will be plotted for a given sampling time only if 2/3 of the individual data at the time point have quantifiable measurements that are within the sampling time window specified in the protocol or ± 10%. An average concentration estimated with less than 2/3 but more than 3 data points may be displayed on the mean concentration plot if determined to be appropriate and will be documented within the final study report.

# Treatment of Outliers during Pharmacokinetic Analysis

Application of this procedure to all PK analyses is not a requirement. Rather, this procedure provides justification for exclusion of data when scientifically appropriate. This procedure describes the methodology for identifying an individual value as an outlier for potential exclusion, but does not require that the value be excluded from analysis. The following methodology will not be used to exclude complete profiles from analysis.

#### Data within an Individual Profile

A value within an individual profile may be excluded from analysis if any of the following criteria are met:

- For PK profiles during multiple dosing, the concentration of the pre-dose sample exceeds all measured concentrations for that individual in the subsequent post-dose samples.
- For PK profiles during single dosing of non-endogenous compounds, the concentration in a pre-dose sample is quantifiable.
- For any questionable datum that does not satisfy the above criteria, the profile will be evaluated and results reported with and without the suspected datum.

#### Data between Individual Profiles

1. If n<6, then the dataset is too small to conduct a reliable range test. Data will be analyzed with and without the atypical value, and both sets of results will be reported.

Final, 28 August 2020 

- 2. If n≥6, then an objective outlier test will be used to compare the atypical value to other values included in that calculation:
  - a. Transform all values in the calculation to the logarithmic domain.
  - b. Find the most extreme value from the arithmetic mean of the log transformed values and exclude that value from the dataset.
  - c. Calculate the lower and upper bounds of the range defined by the arithmetic mean  $\pm 3*SD$  of the remaining log-transformed values.
  - d. If the extreme value is within the range of arithmetic mean  $\pm 3*SD$ , then it is not an outlier and will be retained in the dataset.
  - e. If the extreme value is outside the range of arithmetic mean  $\pm 3*SD$ , then it is an outlier and will be excluded from analysis.

If the remaining dataset contains another atypical datum suspected to be an outlier and  $n \ge 6$  following the exclusion, then repeat step 2 above. This evaluation may be repeated as many times as necessary, excluding only one suspected outlier in each iteration, until all data remaining in the dataset fall within the range of arithmetic mean  $\pm 3*SD$  of the log-transformed values.

# Reporting of Excluded Values

Individual values excluded as outliers will be documented in the final report. Approval of the final report will connote approval of the exclusion.

# 9.3.2 Pharmacokinetic Statistical Methodology

All tests of treatment effects will be conducted at a 2-sided alpha level of 0.1, unless otherwise stated, and all CIs will be given at a 2-sided 90% level.

The primary parameters for analysis will be AUC(0- $\infty$ ) of LY3819253 following SC administration. Other noncompartmental parameters, such as half-life,  $t_{max}$ , apparent clearance, and volume of distribution following SC administration may be reported.

The natural log (ln)-transformed AUC( $0-\infty$ ) will be analyzed using an analysis of variance model. The model will include dose as a factor. Body weight may be tested as a covariate and kept if needed.

The least squares mean for each treatment, difference in least square means between the treatments, and corresponding 90% CI will be calculated; these values will then be back-transformed to give the geometric least square mean, ratio of geometric least square means, and corresponding 90% CI.

Final, 28 August 2020 

# Example SAS code for the analysis:

```
proc mixed data=pk;
  class dose;
  model log_pk = dose / alpha=0.1 cl residual ddfm=kr2;
  lsmeans dose / cl pdiff;
  ods output lsmeans=lsm;
  ods output diffs=diff;
  ods output tests3=tests;
run;
```

In addition to noncompartmental analysis, the data may be combined with data from other studies to be analyzed using non-linear mixed-effect modelling of the PK data. This analysis will be the responsibility of Eli Lilly PK/PD group.

# 9.4 Safety and Tolerability Assessments

#### 9.4.1 Adverse events

Where changes in severity are recorded in the Case Report Form (CRF), each separate severity of the AE will be reported in the listings, only the most severe will be used in the summary tables. A pre-existing condition is defined as an AE that starts before the subject has provided written informed consent and is ongoing at consent. A non-treatment emergent AE is defined as an AE which starts after informed consent but prior to dosing. A TEAE is defined as an AE which occurs postdose or which is present prior to dosing and becomes more severe postdose.

All AEs will be listed. All TEAEs will be summarized by treatment, severity and relationship to the study drug. The frequency (the number of AEs, the number of subjects experiencing an AE and the percentage of subjects experiencing an AE) of TEAEs will be summarized by treatment, Medical Dictionary for Regulatory Activities (MedDRA) version 23.0 system organ class and preferred term. The summary and frequency AE tables will be presented for all causalities and those considered related to the study drug by the investigator. Any SAEs will be listed.

Discontinuations due to AEs will be listed.

#### 9.4.2 Concomitant medication

Concomitant medication will be coded using the WHO drug dictionary (Version March 2020 B3). Concomitant medication will be listed.

# 9.4.3 Clinical laboratory parameters

All clinical chemistry and hematology data will be summarized by parameter and treatment, together with changes from baseline, and listed. Baseline is defined as the Day -1 predose assessment. Urinalysis data will be listed. Additionally, clinical chemistry, hematology and urinalysis data outside the reference ranges will be listed and flagged on individual subject data listings.

Data from SARS-CoV-2 clinical screening, serology, and point-of-care test will be listed, if available.

Final, 28 August 2020 

# 9.4.4 Vital signs

Vital signs data will be summarized by treatment together with changes from baseline, where baseline is defined as the Day 1 predose assessment. Figures of mean vital signs and mean changes from baseline profiles will be presented by treatment.

Values for individual subjects will be listed.

# 9.4.5 Electrocardiogram (ECG)

ECGs will be performed for safety monitoring purposes only and will not be presented. Any clinically significant findings from ECGs will be reported as an AE.

# 9.4.6 Immunogenicity Assessments

The frequency and percentage of subjects with pre-existing antidrug antibody (ADA) and with TE ADAs to LY3819253 will be tabulated and listed only if the data is available.

The frequency and percentage of subjects with cross-reactive and neutralizing antibodies, if measured, may also be tabulated for subjects with TE ADA.

# 9.4.7 Injection-Site Reactions

ISR data (including erythema, induration, pain, pruritus, and edema) will be listed and summarized by treatment in frequency tables. ISR will be listed and may be summarized if there are ≥3 subjects with ISR per dose.

# 9.4.8 Visual Analog Scale (VAS) Analysis

The VAS is a well-validated tool to assess injection site pain; it is presented as a 100 mm line anchored by verbal descriptors, usually "no pain" and "worst imaginable pain." The participant will be asked to rate any pain at the injection site on a scale of 0 to 100 on the line, as soon as possible following each injection.

The data will be listed and summarized by treatment and time point.

# 9.4.9 Hypersensitivity reactions

For all drug hypersensitivity reactions that occur, additional follow-up data will be collected to assess the patient's medical history, alternative causes, and symptoms.

These data will be listed.

#### 9.4.10 Other assessments

All other safety assessments not detailed in this section will be listed but not summarized or statistically analyzed.

Final, 28 August 2020 

# 9.4.11 Safety and Tolerability Statistical Methodology

No inferential statistical analyses are planned.

#### 10. INTERIM ANALYSES

No interim statistical analyses are planned.

# 11. CHANGES FROM THE PROTOCOL SPECIFIED STATISTICAL ANALYSES

There were no changes from the protocol specified statistical analyses.

#### 12. REFERENCES

- 1. International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use, ICH Harmonized Tripartite Guideline, Statistical Principles for Clinical Trials (E9), 5 February 1998.
- 2. International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use, ICH Harmonized Tripartite Guideline, Structure and Content of Clinical Study Reports (E3), 30 November 1995.

#### 13. DATA PRESENTATION

#### 13.1 Derived Parameters

Individual derived parameters (e.g. PK parameters) and appropriate summary statistics will be reported to three significant figures. Observed concentration data, e.g. C<sub>max</sub>, should be reported as received. Observed time data, e.g. t<sub>max</sub>, should be reported as received. N and percentage values should be reported as whole numbers. Median values should be treated as an observed parameter and reported to the same number of decimal places as minimum and maximum values.

# 13.2 Missing Data

Missing data will not be displayed in listings.

# 13.3 Insufficient Data for Presentation

Some of the TFLs may not have sufficient numbers of subjects or data for presentation. If this occurs, the blank TFL shell will be presented with a message printed in the center of the table, such as, "No serious adverse events occurred for this study."

Final, 28 August 2020 

#### Leo Document ID = 9dd5bad7-ce9f-410f-83e3-71987d96ac73

Approver: PPD

Approval Date & Time: 28-Aug-2020 16:17:08 GMT

Signature meaning: Approved

Approver: PPD

Approval Date & Time: 28-Aug-2020 16:31:40 GMT

Signature meaning: Approved

Approver: PPD

Approval Date & Time: 28-Aug-2020 16:44:39 GMT

Signature meaning: Approved

Approver: PPD

Approval Date & Time: 01-Sep-2020 14:56:21 GMT

Signature meaning: Approved